CLINICAL TRIAL: NCT01339377
Title: A Pilot Study to Evaluate the Safety and Effectiveness of Ozone Generated and Injected by the AO-1000 Device in the Treatment of Contained Herniated Discs
Brief Title: Safety and Effectiveness Study of the AO-1000 Device to Treat Contained Herniated Discs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ActiveO Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT2-IPP-001-AO
Record Dates: First submitted 2011-04-19; First posted 2011-04-20 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Disk, Herniated
Keywords: Ozone; Oxygen; Oxygen-Ozone; AO-1000; ActiveO; Herniated Disc; Disc; Lumbar
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AO-1000 Treatment (Experimental): Oxygen-ozone treatment with the AO-1000 device
  Interventions: Device: AO-1000

INTERVENTIONS:
Device: AO-1000 — Mixture of 2 weight% ozone in 98 weight% oxygen injected into the nucleus pulposus of a contained herniated disc.

SUMMARY:
To evaluate the safety and effectiveness of the AO-1000 device to treat and relieve the pain of symptomatic subjects with contained herniated discs. This single-arm pilot study will be used as a go vs. no-go decision on performing a randomized-controlled trial.

The study's primary effectiveness objective is to demonstrate that the patient's functionality (based on Oswestry Disability Index scores) has improved from baseline at one month. The study's primary safety objective is to demonstrate that serious device/procedure related adverse events and subsequent surgical interventions are no greater than those in a literature control of other percutaneous disc decompression procedures at discharge, 1 month, 6 months, and 12 months post-treatment.

Secondary objectives are to demonstrate procedural success and improvement in the pain and function of the subjects at 1, 6, and 12 months using the VAS and ODI scales as well as tracking analgesic medication use. Pain and function scores for each follow-up time will be compared to the baseline scores.

DETAILED DESCRIPTION:
The AO-1000 device provides an oxygen-ozone treatment for contained herniated discs. An oxygen-ozone treatment is a minimally invasive injection for treating disc herniations that is widely practiced in Europe and Asia. This treatment involves the injection of an oxygen-ozone mixture into the herniated disc and/or the paravertebral muscle surrounding the disc. However, there are no medical ozone generators for this procedure that are currently cleared by the FDA for use in the US. Many studies using a wide range of inclusion/exclusion criteria, ozone concentrations, and procedures have been performed to determine the effectiveness of oxygen-ozone treatment.

A meta-analysis of nearly 8,000 patients from published studies shows a mean improvement of 39 mm for VAS and 25.7 for ODI. The likelihood of complications was 0.064%. Furthermore, no cases of discitis were reported after oxygen-ozone therapy, which is unlike all the other methods of disc volume reduction. This is most likely due to the fact that ozone is a strong oxidizer and an excellent disinfecting agent. The complications shown in the meta-analysis were minor and transient, and easily avoidable by utilizing a device such as the AO-1000 that is designed to eliminate these types of complications (ozone leakage into the treatment room and high ozone concentrations) during this procedure. The estimated complication rate from the meta-analysis is consistent with the Italian Oxygen-Ozone Therapy Federation (FIO) results (no procedure-related adverse events in treatments on 15,000 patients).

The safety of the direct injection of oxygen-ozone gas mixture into the nucleus pulposus was well established in these studies. Therefore, the intent of this study is to obtain data to confirm that a 2 weight percent (wt%) oxygen-ozone mixture delivered from the AO-1000 device is safe and effective for the intended use. This clinical study is designed to bridge the AO-1000 to the extensive prior oxygen-ozone treatment safety and effectiveness data between studies such as those found in the Meta-analysis that did not use the AO-1000 as the delivery system.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age
* Herniated disc between L1 and S1 evident on diagnostic imaging
* Sciatica with or without lower back pain for > 3 months
* Failure to improve with non-operative care (Conservative treatment failure)
* Sciatica with or without lower back pain exacerbated by sitting and/or standing with recumbent relief
* A preoperative leg or back VAS (pain) score between 40 and 90 mm on a 100 mm scale. (moderate to severe pain)
* A preoperative ODI (function) score between 40 and 90 (moderate to severe functional disability)
* Able and willing to return for the follow-up evaluations
* The pain must be consistent with the dermatome pattern and must be clearly identifiable to the herniated disc.

Exclusion Criteria:

* Functional neurological deficit evident during neurological exam
* Previous spine surgery in the lumbar region or adjacent to the disc of interest
* Cord compression or cauda equine syndrome
* Structural deformities (e.g. spondylolisthesis, greater than a mild degree of non-discogenic vertebral canal stenosis, greater than a mild degree of scoliosis, spinal fracture, disc herniations > 4 mm, sequestered herniation)
* Extruded/free disc fragment
* Calcified disc fragment
* Disc height loss > 75%
* Inaccessible disc due to, for example, overlap of the iliac wings, and/or steep angulation of the L5/S1 disc space
* Coagulopathy evident on blood sample testing
* Platelet count < 50,000
* International Normalized Ratio (INR) > 1.4
* Partial Thromboplastin Time (PTT) > 1.3
* White blood cell count (WBCC) > 12,000
* Infection as evidenced by subject clinical evaluation, history, and blood test
* Any evidence of osteomyelitis/discitis at any level
* Uncontrolled/acute illness
* Women who are pregnant
* Worker's compensation, injury litigation, disability remuneration
* Participation in another clinical investigation or course of care that may confound the outcome of this study
* Smoker

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint: Change from Baseline ODI Score at 1 Month | 1 month post-treatment
  Mean change from baseline ODI score, analyzed at 1 month. The endpoint will be deemed successful if the mean improvement is statistically shown (p<0.05) to be at least 15 points (the minimum detectable change of the ODI).
Primary Safety Endpoint: Frequency of Serious Adverse Events Compared to Literature Control | 12 months post-treatment
  The endpoint will be deemed successful if the number of serious device/procedure related adverse events are statistically shown (p<0.05) to be no greater than those in a literature control of other percutaneous disc decompression procedures.

SECONDARY OUTCOMES:
Functional improvement | 6 and 12 months post-treatment
  Mean change from baseline ODI score, analyzed at 6 and 12 months. Each endpoint will be deemed successful if the mean improvement is statistically shown (p<0.05) to be at least 15 points (the minimum detectable change of the ODI).
Leg and Back Pain Improvement | 1, 6, and 12 months post-treatment
  Mean change from separate leg and back pain baseline Visual Analog Scale (VAS) scores, analyzed at 1, 6, and 12 months. Each endpoint (leg VAS and back VAS at each follow-up time) will be deemed successful if the mean improvement is statistically shown (p<0.05) to be at least 20 mm (the minimum clinically important difference of the VAS).
Procedural Success | Time of Treatment
  Technical success, as assessed by successful injection of oxygen-ozone mixture confirmed via CT scan performed immediately following the treatment. A treatment will be considered a success if the CT scan shows gas within the target disc.
Analgesic Medication Use | 1, 6, and 12 months post-treatment
  Change in prescription and over-the-counter (OTC) analgesic medication use, including non-steroidal anti-inflammatory drugs (NSAIDs) from baseline, analyzed at 1, 6, and 12 months. Endpoint will be deemed successful if the number of patients using analgesic medication decreases from baseline.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Vancouver General Hospital, Vancouver, British Columbia
  - University of Western Ontario - London Health Sciences Centre, London, Ontario
  - Toronto Western Hospital, Toronto, Ontario

REFERENCES:
- [Background] Steppan J, Meaders T, Muto M, Murphy KJ. A metaanalysis of the effectiveness and safety of ozone treatments for herniated lumbar discs. J Vasc Interv Radiol. 2010 Apr;21(4):534-48. doi: 10.1016/j.jvir.2009.12.393. Epub 2010 Feb 25. PMID 20188591
- [Background] Pellicanò G, Martinelli F, Tavanti V, et al. The Italian Oxygen-Ozone Therapy Federation (FIO) Study on Oxygen-Ozone Treatment of Herniated Disc. Int J Ozone Ther 6:7-15, 2007.
- [Background] Oder B, Loewe M, Reisegger M, Lang W, Ilias W, Thurnher SA. CT-guided ozone/steroid therapy for the treatment of degenerative spinal disease--effect of age, gender, disc pathology and multi-segmental changes. Neuroradiology. 2008 Sep;50(9):777-85. doi: 10.1007/s00234-008-0398-2. Epub 2008 May 16. PMID 18483728
- [Background] Mixter WJ, Barr JS. Rupture of the intervertebral disc with involvement of the spinal canal. N Engl J Med 211:210-215, 1934.
- [Background] Andreula CF, Simonetti L, De Santis F, Agati R, Ricci R, Leonardi M. Minimally invasive oxygen-ozone therapy for lumbar disk herniation. AJNR Am J Neuroradiol. 2003 May;24(5):996-1000. PMID 12748111
- [Background] Andreula C, Muto M, Leonardi M. Interventional spinal procedures. Eur J Radiol. 2004 May;50(2):112-9. doi: 10.1016/j.ejrad.2003.10.013. PMID 15081127
- [Background] Bonetti M, Fontana A, Cotticelli B, Volta GD, Guindani M, Leonardi M. Intraforaminal O(2)-O(3) versus periradicular steroidal infiltrations in lower back pain: randomized controlled study. AJNR Am J Neuroradiol. 2005 May;26(5):996-1000. PMID 15891150
- [Background] Gallucci M, Limbucci N, Zugaro L, Barile A, Stavroulis E, Ricci A, Galzio R, Masciocchi C. Sciatica: treatment with intradiscal and intraforaminal injections of steroid and oxygen-ozone versus steroid only. Radiology. 2007 Mar;242(3):907-13. doi: 10.1148/radiol.2423051934. Epub 2007 Jan 5. PMID 17209164